CLINICAL TRIAL: NCT02667548
Title: Prospective Evaluation of Prognosis of Pci Patients Using Network Data in SHengjing Hospital of China Medical University
Brief Title: Prospective Evaluation of Prognosis of Pci Patients Using Network Data in SHengjing Hospital
Acronym: P-PUSH
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, YU Tong-tong, attending physician, Shengjing Hospital
Other Study IDs: 2016PS04K02
Record Dates: First submitted 2016-01-21; First posted 2016-01-29 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Coronary Heart Disease
Keywords: percutaneous coronary intervention
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A venous blood sample of 10mL will be collected before discharge for biomarker analysis and storage for future genetic studies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients receiving PCI: patients receiving PCI
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — percutaneous coronary intervention

SUMMARY:
Coronary heart disease (CHD) has a serious health threaten to population. PCI is a well-proved measure in CHD management. However, the knowledge about the real-life PCI use and how evidence-based therapies in routine clinical practice is limited. By consecutively recruiting PCI patients in a large-scale hospital in in Northeast China,this study will examine various real-life factors, that may affect patients recovery after the procedure. Practical guidelines, appropriateness criteria and quality evaluative system for PCI will be established based on the findings, to improve patients outcomes in future finally.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a major concern in public health in China. Relatively limited information is available about how evidence-based therapies are incorporated appropriately into routine clinical practice. Practical and applied knowledge from large unselected population is needed to guide practice for quality improvement.

This study will enroll patients undergoing PCI in a large-scale hospital in in Northeast China. At study entry, participants will be interviewed during their index hospitalization, to collect information about symptoms, functioning, quality of life, and medical care. Demographic characteristics, medical history, clinical features, diagnostic tests, medications, procedures, and in-hospital outcomes of patients will be abstracted from medical records by well trained professional abstractors. CAG imaging will be reviewed by 2 cardiologists through PACS. Other Procedural data, including stent type, total stent length and so on, came from operation records of PCI cases finished by operators. At 1 month, 6 month, 12 month, 3 year and 5 year after discharge, participants will return to the clinic for follow up visits, a face-to-face interview will be conducted to get information about clinical events, symptoms, functioning, quality of life, and medical care during the recovery period. If participants can not return to the clinic for follow up visits,a telephone interview will be conducted to get the related information. Before discharge,, blood sample will be collected. Participants' blood samples will be stored for future biologic and genetic studies. This study will examine various real-life factors that may affect patients recovery after PCI, including patients' characteristics and treatment measures. Practical guidelines, quality evaluative system, and appropriateness criteria will be established based on the findings, to improve patients outcomes in future finally.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients undergoing a percutaneous coronary intervention (PCI) for coronary lesions.

Exclusion Criteria:

* Previously enrolled in the R-PUSH study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In department of Cardiology,Shengjing Hospital of China Medical University, 7000 hospitalized patients undergoing Percutaneous Coronary Intervention will be enrolled consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2016-01; Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Major adverse cardiovascular events (MACE) | 5 year
  Composite of major adverse cardiovascular events (MACE) including cardiac death, non-fatal AMI, coronary revascularization procedure, or ischemic stroke

SECONDARY OUTCOMES:
Percentage of Participants with all-cause death | 5 year
Percentage of Participants with cardiac death | 5 year
Percentage of Participants with non-fatal AMI | 5 year
Percentage of Participants with coronary revascularization procedure | 5 year
  coronary revascularization procedure includs any unplanned repeat PCI or surgical bypass of target or non-target vessels.
Percentage of Participants with ischemic stroke | 5 year
Percentage of Participants with Cardiac Re-admission | 5 year
  Cardiac Re-admission includes any re-admission because of aggravation of heart failure or angia.
Percentage of Participants with Adherence to medications for secondary prevention | 5 year
  Taking the following medications for 6 or more days per week: aspirin, clopidogrel, ACEI/ARB, statin and beta-blockers
Number of Participants who quit smoking | 5 year
Symptoms status as assessed by SAQ | 5 year
Quality of life as assessed by EQ-5D | 5 year
Depression as assessed by PHQ-8 | 5 year
Stress as assessed by PSS-4 | 5 year

OTHER OUTCOMES:
Cognitive function as assessed by MMSE | 5 year
Sexual activity as assessed by a question: Have participants had sex or sexual activity since participants were hospitalized for heart attack or heart problem? Response Options:Dichotomous (Y/N) | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Tongtong Yu, Doctor, Principal Investigator — Shengjing Hospital

IPD SHARING:
Plan to Share IPD: No
We will not share IPD to protect our data very well.